CLINICAL TRIAL: NCT05904977
Title: Preliminary Study on the Metastatic Rate and Clinical Significance of the Anterior Leaf of Vesicouterine Ligament in Early Stage Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-446-01
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; Radical hysterectomy; Ultrastaging; Vesicouterine ligament
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type B resection: The patients reviced type B resection of the antierior leaf of vesicouterine ligament
  Interventions: Procedure: Type B resection or type C resection of the anterior leaf of vesicouterine ligament during the radical hysterectomy (type C)
- Type C resection: The patients reviced type C resection of the antierior leaf of vesicouterine ligament
  Interventions: Procedure: Type B resection or type C resection of the anterior leaf of vesicouterine ligament during the radical hysterectomy (type C)

INTERVENTIONS:
Procedure: Type B resection or type C resection of the anterior leaf of vesicouterine ligament during the radical hysterectomy (type C) — The patients with cervical cancer who underwent abdominal radical hysterectomy（type C）plus pelvic lymph node dissection by the same surgical team at the Department of Gynecological Oncology, Sun Yat-sen Memorial Hospital, Sun Yat-Sen University, were included. According to the resection range of the anterior leaf of vesicouterine ligament (VUL), patients were divided into type C resection group (near the bladder wall) and B type resection group (above the ureter).

SUMMARY:
The purpose of this study is to preliminarily explore the metastatic rate and clinical significance of the anterior leaf of vesicouterine ligament resection for early stage cervical cancer, so as to further improve the postoperative quality of life of patients and reduce the incidence of postoperative urinary complications.

DETAILED DESCRIPTION:
The patients with cervical cancer who underwent abdominal radical hysterectomy（type C）plus pelvic lymph node dissection by the same surgical team at the Department of Gynecological Oncology, Sun Yat-sen Memorial Hospital, Sun Yat-Sen University, were included. According to the resection range of the anterior leaf of vesicouterine ligament (VUL), patients were divided into type C resection group (near the bladder wall) and B type resection group (above the ureter). The anterior leaf of the VUL in the type C resection group was sent to pathological biopsy separately, and the metastasis rate was further clarified by the pathological "ultrastaging" method. By comparing the clinicopathological characteristics of patients with metastasis and non-metastasis, the potential risk factors of VUL metastasis were analyzed. The oncological outcomes of patients with different resection range of the anterior VUL were compared. At the same time, the Functional Assessment of Cancer Therapy-Cervical（FACT-Cx）cervical cancer patient quality of life score table was used to evaluate cervical cancer patients after surgery. The relevant factors that may affect the quality of life score are included in the multiple linear regression analysis to obtain independent risk factors that affect the quality of life of the patient after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of squamous, adenocarcinoma, or adenosquamous cervical carcinoma (even neuroendocrine or clear cell carcinoma)
2. Radiographically confirmed tumor limited to the cervix or upper third vagina, but without evidence of lymph node metastasis
3. Stage IA2-IIA2 ( FIGO 2018)
4. Treated initially or just underwent cervical conization before
5. Underwent the abdominal type C (Q-M classification) radical hysterectomy with pelvic lymph node dissection by the same team
6. Underwent the bilateral type C AL-VUL resection during the surgery
7. The Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

1. Not stage IA2-IIA2 ( FIGO 2018)
2. History of abdominal or pelvic radiotherapy
3. Evidence of metastatic disease detected by PECT, MRI or CT
4. The surgeon evaluated the patient as unsuitable for abdominal radical hysterectomy or the patient as refusing abdominal surgery
5. Patients with other mailgnant tumors except cervical cancer
6. Incompetence of the clinical, surgical and pathological data

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with cervical cancer who underwent abdominal radical hysterectomy（type C）plus pelvic lymph node dissection by the same surgical team at the Department of Gynecological Oncology, Sun Yat-sen Memorial Hospital, Sun Yat-Sen University, were included. According to the resection range of the anterior leaf of vesicouterine ligament (VUL), patients were divided into type C resection group (near the bladder wall) and B type resection group (above the ureter).
Sampling Method: Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Metastatic rate of the anterior leaf of vesicouterine ligament | 1 year (Postoperative pathological confirmation date)
  The metastasis rate of anterior leaf of VUL (%) = (case number of positive metastatic lesion detected by H&E staining + case number of positive metastatic lesion diagnosed by "ultrastaging") / Total number of the patients with cervical cancer who underwent abdominal radical hysterectomy（type C）plus pelvic lymph node dissection by the samesurgical team ×100%

SECONDARY OUTCOMES:
Incidence of postoperative adjuvant therapy in patients with metastasis in the anterior leaf of VUL | 1 year after surgery
  Clinical data
Incidence of postoperative urinary dysfunction in two groups | 1 year after surgery
  Follow-up and subjective description
Postoperative quality of life scores in two groups | 1，2，3 years after surgery
  The Functional Assessment of Cancer Therapy-Cervical（FACT-Cx）cervical cancer patient quality of life score table
DFS | 3 years after surgery
  Disease-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Huaiwu Lu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arbyn M, Weiderpass E, Bruni L, de Sanjose S, Saraiya M, Ferlay J, Bray F. Estimates of incidence and mortality of cervical cancer in 2018: a worldwide analysis. Lancet Glob Health. 2020 Feb;8(2):e191-e203. doi: 10.1016/S2214-109X(19)30482-6. Epub 2019 Dec 4. PMID 31812369
- [Background] Cao TT, Wen HW, Gao YN, Lyu QB, Liu HX, Wang S, Wang SY, Sun HX, Yu N, Wang HB, Li Y, Wang ZQ, Chang OH, Sun XL, Wang JL. Urodynamic assessment of bladder storage function after radical hysterectomy for cervical cancer. Chin Med J (Engl). 2020 Oct 5;133(19):2274-2280. doi: 10.1097/CM9.0000000000001014. PMID 32925291
- [Background] Querleu D, Cibula D, Abu-Rustum NR. 2017 Update on the Querleu-Morrow Classification of Radical Hysterectomy. Ann Surg Oncol. 2017 Oct;24(11):3406-3412. doi: 10.1245/s10434-017-6031-z. Epub 2017 Aug 7. PMID 28785898
- [Background] Kim CH, Soslow RA, Park KJ, Barber EL, Khoury-Collado F, Barlin JN, Sonoda Y, Hensley ML, Barakat RR, Abu-Rustum NR. Pathologic ultrastaging improves micrometastasis detection in sentinel lymph nodes during endometrial cancer staging. Int J Gynecol Cancer. 2013 Jun;23(5):964-70. doi: 10.1097/IGC.0b013e3182954da8. PMID 23694985
- [Background] Zand B, Euscher ED, Soliman PT, Schmeler KM, Coleman RL, Frumovitz M, Jhingran A, Ramondetta LM, Ramirez PT. Rate of para-aortic lymph node micrometastasis in patients with locally advanced cervical cancer. Gynecol Oncol. 2010 Dec;119(3):422-5. doi: 10.1016/j.ygyno.2010.08.012. Epub 2010 Sep 15. PMID 20837355
- [Background] Kornblith AB, Huang HQ, Walker JL, Spirtos NM, Rotmensch J, Cella D. Quality of life of patients with endometrial cancer undergoing laparoscopic international federation of gynecology and obstetrics staging compared with laparotomy: a Gynecologic Oncology Group study. J Clin Oncol. 2009 Nov 10;27(32):5337-42. doi: 10.1200/JCO.2009.22.3529. Epub 2009 Oct 5. PMID 19805678
- [Background] Narayansingh GV, Miller ID, Sharma M, Welch CJ, Sharp L, Parkin DE, Cruickshank ME. The prognostic significance of micrometastases in node-negative squamous cell carcinoma of the vulva. Br J Cancer. 2005 Jan 31;92(2):222-4. doi: 10.1038/sj.bjc.6602343. PMID 15655537